CLINICAL TRIAL: NCT01093196
Title: A Phase 3, Intergroup Multicentre, Randomized, Controlled 3 Arm Parallel Group Study to Determine the Efficacy and Safety of Lenalidomide in Combination With Dexamethasone (RD) Versus Melphalan, Prednisone and Lenalidomide (MPR) Versus Cyclophosphamide, Prednisone and Lenalidomide (CPR) in Newly Diagnosed Elderly Multiple Myeloma Subjects
Brief Title: Lenalidomide and Dexamethasone Versus Melphalan Prednisone and Lenalidomide Versus Cyclophosphamide, Prednisone and Lenalidomide in Elderly Multiple Myeloma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMN01
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Elderly Patients; Diagnosis; Lenalidomide; Prednisone; Melphalan; Dexamethasone; Cyclophosphamide
MeSH Terms: conditions — Multiple Myeloma; Disease | interventions — Melphalan; Prednisone; Lenalidomide; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rd (Active Comparator): Induction treatment with oral Lenalidomide and low dose dexamethasone followed by maintenance therapy with Lenalidomide alone or Lenalidomide and Prednisone
  Interventions: Drug: Lenalidomide, dexamethasone
- MPR (Experimental): Induction treatment with oral Lenalidomide, Prednisone and Melphalan followed by maintenance therapy with Lenalidomide alone or Lenalidomide and Prednisone
  Interventions: Drug: Melphalan, Prednisone, Lenalidomide
- CPR (Experimental): Induction treatment with oral Lenalidomide, Cyclophosphamide and Prednisone for followed by maintenance therapy with Lenalidomide alone or Lenalidomide and Prednisone.
  Interventions: Drug: Cyclophosphamide, Prednisone, Lenalidomide

INTERVENTIONS:
Drug: Melphalan, Prednisone, Lenalidomide — Induction: 9 courses every 28 days - oral Lenalidomide for 21 days followed by a 7 days rest period; oral Melphalan for 4 days, followed by a 24 days rest period [different doses according to the age of patients (65-75 or >75 years old);oral Prednisone for 4 days followed by a 24 day rest period.
  Maintenance: ARM A1, B1 and C1 - oral Lenalidomide on day 1-21 followed by a 7 days rest period.
  ARM A2,B2 and C2:oral Lenalidomide on day 1-21 followed by a 7 days rest period and oral Prednisone every other day.Each cycle will be repeated every 28 days, until any sign of disease progression(PD).
  Arms: MPR
Drug: Cyclophosphamide, Prednisone, Lenalidomide — Induction: 9 cycles every 28 days:Lenalidomide will be given orally at the dose of 25 mg/day for 21 days followed by a 7 days rest period (day 22 to 28;Cyclophosphamide will be given orally at the dose of 50 mg /day for 21 days followed by a 7 day rest period (days 1 to 28) in patients 65-75 years old and 50 mg every other day (days 1 to 20 followed by a 8 days rest period [day 21 to 28]) in patients older than 75 years.Prednisone will be given orally at the dose of 25 mg every other day (days 1 to 28.Each cycle will be repeated every 28 days, until any sign of disease progression(PD).
  Arms: CPR
Drug: Lenalidomide, dexamethasone — Induction: 9 course every 28 days-Lenalidomide will be given orally at the dose of 25 mg/day for 21 days followed by a 7 days rest period (day 22 to 28); Dexamethasone will be given orally at the dose of 40 mg on days 1, 8, 15 and 22 every 28 days in patients 65-75 years old and at the dose of 20 mg on days 1,8,15 and 22 every 28 days in patients older than 75 years. Maintenance:After 2-3 months from the completion of the last induction cycle, patients will start maintenance therapy according to physician willing and general dose-reduction rules.ARM A1, B1 and C1:Lenalidomide will be given at the dose of 10 mg/day on day 1-21 followed by a 7 days rest period. ARM A2, B2 and C2:Lenalidomide will be given at the dose of 10 mg/day on day 1-21 followed by a 7 days rest period; Prednisone will be given orally at the dose of 25 mg every other day (days 1 to 28) Each cycle will be repeated every 28 days, until any sign of disease progression (PD).
  Arms: Rd

SUMMARY:
This is a multicenter, randomized, controlled, 3 arm parallel group study designed to evaluate the efficacy and safety of three all-oral combinations: lenalidomide with dexamethasone (Rd) in comparison with lenalidomide in association with MP (MPR) and lenalidomide in association with cyclophosphamide - prednisone (CPR) in newly diagnosed symptomatic MM patients. This protocol also provides a substudy designed to observe asymptomatic patients excluded to the protocol that in any case could be inserted in the study.

DETAILED DESCRIPTION:
This is an intergroup multicenter, randomized, open label study designed to compare the efficacy and safety of Rd with MPR and CPR in newly diagnosed symptomatic MM patients who are 65 years of age or older. Potential study subjects will sign an informed consent prior to undergoing any study related procedure.

This study consists of 3 phases for each study subject: Pre-treatment, Treatment and Follow up.Pre-treatment period: patients will undergo screening for protocol eligibility within 28 days (4weeks) prior to randomization.

Subjects who meet all the inclusion criteria will be randomized based on a computer-generated randomization schedule prepared by the Coordinating Centre. The first randomization will occur for the induction treatment: Arm A (Rd) or B (MPR) or C (CPR). Within each arm patients will be then randomized for the maintenance treatment(lenalidomide or lenalidomide and prednisone): Arms A1 (R) and A2 (RP); Arms B1 (R) and B2 (RP); Arms C1 (R) and C2 (RP). Randomization will be concealed until the end of the induction period for the maintenance treatment. Patients will be stratified at randomization according to the International Staging System (5) and age (< 75 years vs > 75 years).Treatment period includes induction and maintenance. During the induction and maintenance phases, all patients will attend periodic study center visits in order to asses the safety and efficacy of the treatment. This protocol also provides a substudy designed to observe asymptomatic patients excluded to the protocol that in any case could be inserted in the study . The asymptomatic patient is characterized by the absence of end-organ damage or tissue involvement, such as anemia, bone lesions, hypercalcemia, and renal failure, or by other relevant clinical conditions, such as hyperviscosity, amyloidosis, and recurrent infections (CRAB).

ELIGIBILITY:
Inclusion Criteria:

* Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Patient is 65 years old or older at the time of signing the informed consent or younger patients not candidate to high dose therapy
* Female patient is either post-menopausal or surgically sterilized or, if at child-bearing potential†, must:

  * understand that the study medication could have an expected teratogenic risk
  * Agree to use, and be able to comply with, effective contraception without interruption, 4 weeks before starting study drug, throughout study drug therapy (including dose interruptions) and for 4 weeks after the end of study drug therapy, even if she has amenorrhea. This applies unless the subject commits to absolute and continued abstinence confirmed on a monthly basis. The following are effective methods of contraception*
* Implant**
* Levonorgestrel-releasing intrauterine system (IUS)**
* Medroxyprogesterone acetate depot
* Tubal sterilisation
* Sexual intercourse with a vasectomised male partner only; vasectomy must be confirmed by two negative semen analyses
* Ovulation inhibitory progesterone-only pills (i.e., desogestrel)

Combined oral contraceptive pills are not recommended. If a subject was using combined oral contraception, she must switch to one of the methods above. The increased risk of VTE continues for 4 to 6 weeks after stopping combined oral contraception.

* prophylactic antibiotics should be considered at the time of insertion particularly in patients with neutropenia due to risk of infection

  * Agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 mIU/ml not more than 3 days before the start of study medication once the subject has been on effective contraception for at least 4 weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.
  * Agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization. These tests should be performed not more than 3 days before the start of next treatment. This requirement also applies to women of childbearing potential who practice complete and continued abstinence

    - Male subjects must
  * Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study therapy if their partner is of childbearing potential and has no contraception.
  * Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.

    - All subjects must
  * Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
  * Agree not to share study medication with another person and to return all unused study drug to the investigator.

    - Patient was previously diagnosed with symptomatic MM based on standard criteria, and has measurable disease, defined as follows:
  * Secretory myeloma: any quantifiable serum monoclonal protein value (generally, but not necessarily, greater than 1 g/dL of IgG M-Protein and greater than 0.5 g/dL of IgA M-Protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours;
  * Non-secretory myeloma: > 30% plasma cells in the bone marrow and at least one plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e., MRI or CT scan).

    * Patient has a baseline bone marrow sample available for cytogenetics, that will be processed and eventually centralized within each country.
    * Patient has a Karnofsky performance status _ 60%.
    * Patient has a life-expectancy > 6 months
    * Patients must have a adequate cardiac function
    * Patients must have adequate pulmonary function
    * Patient has the following laboratory values within 14 days before Baseline (day 1 of the Cycle 1):
    * Platelet count ≥ 75 x 109/L without transfusion support within 7 days before the test.
    * Absolute neutrophil count (ANC) ≥1.0 x 109/L without the use of growth factors.
    * Corrected serum calcium ≤14 mg/dL (3.5 mmol/L).
    * Aspartate transaminase (AST): ≤2.5 x the upper limit of normal (ULN).
    * Alanine transaminase (ALT): ≤ 2.5 x the ULN.
    * Total bilirubin: ≤1.5 x the ULN.
    * Calculated or measured creatinine clearance: ≥30 mL/minute

Exclusion Criteria:

* Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid; < to the equivalent of dexamethasone 40 mg/day for 4 days).
* Any serious medical condition, including the presence of laboratory abnormalities, which places the subject at an unacceptable risk if he or she participates in this study or confounds the experimental ability to interpret data from the study.
* Pregnant or lactating females.
* Prior history of malignancies, other than multiple myeloma, unless the subject has been free of the disease for ≥3 years. Exceptions include the following: Basal cell carcinoma of the skin, Squamous cell carcinoma of the skin, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 5 years

SECONDARY OUTCOMES:
Overall Survival | 5 years
Overall Response Rate | 5 years
Time to progression | 5 years
Time and duration of response | 5 years
Time to next therapy | 5 years
Grade 3-4 hematological and non-hematological adverse events (AEs) | 5 years
Prognosis and cytogenetic abnormalities | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mario Boccadoro, MD, Study Chair — Fondazione EMN Italy Onlus
Locations (1):
- Division Of Hematology, A.O.U. Città della Salute e della Scienza di Torino, Torino, TO, Italy

REFERENCES:
- [Derived] Bringhen S, D'Agostino M, Paris L, Ballanti S, Pescosta N, Spada S, Pezzatti S, Grasso M, Rota-Scalabrini D, De Rosa L, Pavone V, Gazzera G, Aquino S, Poggiu M, Santoro A, Gentile M, Baldini L, Petrucci MT, Tosi P, Marasca R, Cellini C, Palumbo A, Falco P, Hajek R, Boccadoro M, Larocca A. Lenalidomide-based induction and maintenance in elderly newly diagnosed multiple myeloma patients: updated results of the EMN01 randomized trial. Haematologica. 2020 Jul;105(7):1937-1947. doi: 10.3324/haematol.2019.226407. Epub 2019 Oct 3. PMID 31582542
- [Derived] Larocca A, Mina R, Offidani M, Liberati AM, Ledda A, Patriarca F, Evangelista A, Spada S, Benevolo G, Oddolo D, Innao V, Cangiolosi C, Bernardini A, Musto P, Amico V, Fraticelli V, Paris L, Giuliani N, Falcone AP, Zambello R, De Paoli L, Romano A, Palumbo A, Montefusco V, Hajek R, Boccadoro M, Bringhen S. First-line therapy with either bortezomib-melphalan-prednisone or lenalidomide-dexamethasone followed by lenalidomide for transplant-ineligible multiple myeloma patients: a pooled analysis of two randomized trials. Haematologica. 2020 Apr;105(4):1074-1080. doi: 10.3324/haematol.2019.220657. Epub 2019 Jun 27. PMID 31248973
- [Derived] Montefusco V, Gay F, Spada S, De Paoli L, Di Raimondo F, Ribolla R, Musolino C, Patriarca F, Musto P, Galieni P, Ballanti S, Nozzoli C, Cascavilla N, Ben-Yehuda D, Nagler A, Hajek R, Offidani M, Liberati AM, Sonneveld P, Cavo M, Corradini P, Boccadoro M. Outcome of paraosseous extra-medullary disease in newly diagnosed multiple myeloma patients treated with new drugs. Haematologica. 2020 Jan;105(1):193-200. doi: 10.3324/haematol.2019.219139. Epub 2019 Jun 20. PMID 31221778
- [Derived] Magarotto V, Bringhen S, Offidani M, Benevolo G, Patriarca F, Mina R, Falcone AP, De Paoli L, Pietrantuono G, Gentili S, Musolino C, Giuliani N, Bernardini A, Conticello C, Pulini S, Ciccone G, Maisnar V, Ruggeri M, Zambello R, Guglielmelli T, Ledda A, Liberati AM, Montefusco V, Hajek R, Boccadoro M, Palumbo A. Triplet vs doublet lenalidomide-containing regimens for the treatment of elderly patients with newly diagnosed multiple myeloma. Blood. 2016 Mar 3;127(9):1102-8. doi: 10.1182/blood-2015-08-662627. Epub 2016 Jan 4. PMID 26729895
- [Derived] Palumbo A, Bringhen S, Mateos MV, Larocca A, Facon T, Kumar SK, Offidani M, McCarthy P, Evangelista A, Lonial S, Zweegman S, Musto P, Terpos E, Belch A, Hajek R, Ludwig H, Stewart AK, Moreau P, Anderson K, Einsele H, Durie BG, Dimopoulos MA, Landgren O, San Miguel JF, Richardson P, Sonneveld P, Rajkumar SV. Geriatric assessment predicts survival and toxicities in elderly myeloma patients: an International Myeloma Working Group report. Blood. 2015 Mar 26;125(13):2068-74. doi: 10.1182/blood-2014-12-615187. Epub 2015 Jan 27. PMID 25628469